CLINICAL TRIAL: NCT02121301
Title: Phase 2, Single-Center, Randomized, Double-Masked, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of SkQ1 Ophth Sol'n in the Environment and During Challenge in the Controlled Adverse Environment (CAE) Model for the Treatment of DES
Brief Title: A Clinical Study to Assess the Safety and Efficacy of an Ophthalmic Solution (SkQ1) in the Treatment of Dry Eye Syndrome (DES)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mitotech, SA (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-110-0006
Record Dates: First submitted 2014-04-17; First posted 2014-04-23 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye; Dry Eye Syndrome; SkQ1; Keratoconjunctivitis; Dry Eye Disease
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes; Keratoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose SkQ1 (Experimental): Drug: Low Dose 0.155µg/mL SkQ1 ophthalmic solution administered twice daily for 28 days
  Interventions: Drug: Low Dose 0.155µg/mL SkQ1 ophthalmic solution
- High Dose SkQ1 (Experimental): Drug: High Dose 1.55µg/mL SkQ1 ophthalmic solution administered twice daily for 28 days
  Interventions: Drug: High Dose 1.55µg/mL SkQ1 ophthalmic solution
- Placebo (vehicle) (Placebo Comparator): Drug: Placebo (vehicle) ophthalmic solution administered twice daily for 28 days
  Interventions: Drug: Placebo (Vehicle) opthalmic solution

INTERVENTIONS:
Drug: Low Dose 0.155µg/mL SkQ1 ophthalmic solution — eyedrops
  Arms: Low Dose SkQ1
Drug: High Dose 1.55µg/mL SkQ1 ophthalmic solution — eyedrops
  Arms: High Dose SkQ1
Drug: Placebo (Vehicle) opthalmic solution — eyedrops
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to evaluate whether SkQ1 ophthalmic solutions are safe and effective compared to placebo for the treatment of the signs and symptoms of dry eye syndrome.

DETAILED DESCRIPTION:
Single-center, double-masked, randomized, placebo-controlled study comprising 4 visits over the course of approximately 5 weeks. The study included a 1-week placebo (SkQ1 vehicle) run-in period between Visit 1 and Visit 2, and approximately 28 days of twice daily (BID) dosing (Visit 2 - Visit 4). Qualified subjects were randomized 1:1:1 to receive either 1.55 µg/mL SkQ1 ophthalmic solution, 0.155 µg/mL SkQ1 ophthalmic solution, or placebo (vehicle of SkQ1 ophthalmic solution).

The following primary endpoints were tested:

* Corneal Fluorescein staining in the inferior region Pre-CAE at Visit 4 (Day 29), as measured by the Ora Calibra Scale in the worst eye at baseline;
* Worst dry eye symptom (ocular discomfort, dryness, or grittiness - as determined from subject diary data recorded during the 1-week run-in period between Visit 1 and Visit 2) evaluated over the seven days preceding Visit 4 (not including day of visit) during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female of any race, at least 18 years of age
* Have provided written informed consent
* Have a reported history of dry eye syndrome
* Have a history of use or desire to use eye drops for dry eye

Exclusion Criteria:

* Have any clinically significant eye findings that require therapeutic treatment or may interfere with study parameters
* Have previously had LASIK surgery within the last 12 months
* Have used Restasis® within 30 days of Visit 1
* Be a woman who is pregnant, nursing or planning a pregnancy
* Be unwilling to submit a urine pregnancy test if of childbearing potential
* Have a known allergy and/or sensitivity to the test article or its components, including the preservative benzalkonium chloride
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Lawrence General Hospital
Locations (1):
- Lawrence General Hospital, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrov A, Perekhvatova N, Skulachev M, Stein L, Ousler G. SkQ1 Ophthalmic Solution for Dry Eye Treatment: Results of a Phase 2 Safety and Efficacy Clinical Study in the Environment and During Challenge in the Controlled Adverse Environment Model. Adv Ther. 2016 Jan;33(1):96-115. doi: 10.1007/s12325-015-0274-5. Epub 2016 Jan 5. PMID 26733410

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose SkQ1: Low Dose 0.155 μg/mL SkQ1 ophthalmic solution
- High Dose SkQ1: High Dose 1.55 μg/mL SkQ1 ophthalmic solution
- Placebo (Vehicle): Placebo (vehicle) ophthalmic solution
Period: Overall Study
Arm/Group | Low Dose SkQ1 | High Dose SkQ1 | Placebo (Vehicle)
Started | 30 | 30 | 31
Completed | 29 | 26 | 30
Not Completed | 1 | 4 | 1
Not completed — Protocol Violation | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Dose - SkQ1: Low Dose 0.155 μg/mL SkQ1 ophthalmic solution
- High Dose - SkQ1: High Dose 1.55 μg/mL SkQ1 ophthalmic solution
- Total: Total of all reporting groups
Arm/Group | Low Dose - SkQ1 | High Dose - SkQ1 | Placebo (Vehicle) | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 10 | 49
  >=65 years | 10 | 11 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.25) | 59.5 (11.69) | 64.6 (9.76) | 62 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 25 | 67
  Male | 9 | 9 | 6 | 24
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 31 | 91

OUTCOME MEASURES:

1. Primary Outcome: Inferior Corneal Fluorescein Staining
Description: The dry eye sign primary efficacy variable of corneal fluorescein staining of the inferior region of the eye measured on a 0-4 point scale where 0 = no staining and 4 = most staining between treatment arms at day 29
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose SkQ1 | High Dose SkQ1 | Placebo (Vehicle)
Number analyzed (Participants) | 30 | 30 | 31
units on a scale | 2.40 (0.675) | 2.07 (0.704) | 2.11 (0.771)

2. Primary Outcome: Worst Symptom Based on Diary Data
Description: Worst dry eye symptom (as determined from subject diary data recorded during the 1-week run-in period) evaluated over the seven days preceding Day 29 during the treatment period. The scale was on a 0-5 range where 0= no symptoms and 5= worst symptoms measured for a number of dry eye symptoms.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose SkQ1 | High Dose SkQ1 | Placebo (Vehicle)
Number analyzed (Participants) | 30 | 30 | 31
units on a scale | 2.54 (0.993) | 2.52 (0.899) | 2.39 (1.063)

ADVERSE EVENTS:
Time Frame: From dilating drop at Day -7 through end of study (Day 29)
Groups:
- Low Dose SkQ1: Low Dose 0.155 µg/mL SkQ1 opthalmic solution
- High Dose SkQ1: High Dose 1.55 µg/mL SkQ1 opthalmic solution
Arm/Group | Low Dose SkQ1 | High Dose SkQ1 | Placebo (Vehicle)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose SkQ1 (N=30) | High Dose SkQ1 (N=30) | Placebo (Vehicle) (N=31)
discomfort (Eye disorders) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect cooperation among all parties involved in the study. Authorship will be established before writing the manuscript. The study sponsor will have the final decision regarding the manuscript and publication.